CLINICAL TRIAL: NCT07378670
Title: Robot-assisted vs. Open Inguinal Lymphadenectomy for Penile Cancer - a Prospective Randomized Trial With a Supporting Translational Program
Brief Title: DEfeating PEnile CAncer-2
Acronym: DEPECA-2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Institut für Klinisch-Onkologische Forschung (IKF) Frankfurt (Unknown)
Responsible Party: Principal Investigator, Igor Tsaur, Univ.-Prof. Dr. med. Igor Tsaur, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEPECA-2
Record Dates: First submitted 2026-01-09; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Penile Cancer; Penile Neoplasms Malignant
Keywords: robotic inguinal lymph node dissection; inguinal lymphadenectomy; surgical outcome
MeSH Terms: conditions — Penile Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- open inguinal lymphadenectomy (Active Comparator)
  Interventions: Procedure: open inguinal lymphadenectomy
- robot-assisted inguinal lymphadenectomy (Experimental)
  Interventions: Procedure: robot-assisted inguinal lymphadenectomy

INTERVENTIONS:
Procedure: open inguinal lymphadenectomy — open inguinal lymphadenectomy
  Arms: open inguinal lymphadenectomy
Procedure: robot-assisted inguinal lymphadenectomy — robot-assisted inguinal lymphadenectomy
  Arms: robot-assisted inguinal lymphadenectomy

SUMMARY:
Open inguinal lymphadenectomy (O-ILAD) is the current standard of care for invasive staging and simultaneously the curative approach for patients with PeCa and elevated risk for or clinically detectable lymphatic disease in the groin. The high rate of complications of this surgical procedure, which are often mutilating and associated with a long-term convalescence, leads to a critical delay in initiation of adjuvant systemic therapy. Being in apprehension of these postsurgical adversities, physicians are often reluctant with indicating this procedure, thus depriving their patients of the vital prognosis-relevant care. In the sum, these obstacles inevitably result in inferior oncologic outcomes. Aiming to decrease postsurgical detrimental sequelae, several attempts to modify radicality of the technique, including inter alia a radioguided approach of sentinel lymph node resection, have been presented in the last decades. Unfortunately, utilization of the sentinel lymph node technique outside of a few highly specialized referral centers is prone to a significant false negativity, while other approaches are associated with inconsistent oncological and perioperative outcomes, hence precluding a general breakthrough in the surgical management of the groin lymph nodes. Thus, a high unmet medical need exists for the establishment of an approach with the lowest possible rate of complications and at the same time the optimal oncological safety.

In this context, preliminary evidence from small sample studies points to a promising potential of minimally invasive surgery to be further tested in the setting of inguinal lymphadenectomy. A recent retrospective single-center report on robot-assisted inguinal lymphadenectomy (R-ILAD) showed that the rate of major complications was only as low as 2%. On the contrary, the rate of major complications in our own and other O-ILAD series was approx. 30%.

DEPECA-2 is a prospective randomized multicenter trial, in which R-ILAD will be tested vs. O-ILAD on the 1b level of evidence for the first time. The scientific value of the project is significantly substantiated by a comprehensive translational research program, which includes inflammatory and oncologic biomarker research, as well as functional validation in preclinical models. The results of this trial will foster further optimization of outcomes in the surgical management of PeCa.

DETAILED DESCRIPTION:
In contrast to the developing world with the incidence of 2.8-6.8 per 100,000 men, penile cancer (PeCa) is an orphan disease in Western countries where the incidence is below 1.0 per 100 000 males (Douglawi-2019). A plethora of risk factors have been identified including lack of neonatal circumcision, phimosis, chronic inflammation, lichen sclerosus, socioeconomic status, obesity, smoking, psoralen UV-A phototherapy, premalignant lesions as well as impaired immune response (Douglawi-2019, Thomas-2020). Moreover, human papilloma virus (HPV) has been attributed to nearly 40-50% of cases (Diorio-2016, Backes-2009). The disease most commonly affects men in their 6th decade of life, whereas young males may be at a higher risk for more aggressive tumor characteristics if diseased (Paiva-2015). PeCa is a distinctly aggressive malignancy characterized by a rapid tumor growth as well as prompt lymphatic metastasis (Hakenberg-2015). Whereas for localized disease cure can be achieved in most patients, prognosis is literally fatal for metastatic PeCa (Thomas-2021). After failing the first-line cisplatin-based chemotherapy providing a progression-free survival of 20 weeks and a response rate of 30%, overall survival falls short of 6 months (Wang-2015). It is a matter of concern that contemporary reports from the USA, France, and Norway have shown that survival of PeCa patients remained unchanged over respective periods of 10, 20, and 60 years despite all efforts in the amelioration of diagnostic and therapeutic paradigms (Daubisse-Marliac-2017, Hansen-2018, Pham-2017). It is furthermore noteworthy that most currently used cytotoxic concepts for this less chemo-responsive condition have been introduced a decade ago at the earliest (Thomas-2021). Besides frequently encountered patient-related issues as delayed medical consultations impairing oncologic outcomes, several other aspects contribute to the lack of progress in the treatment of this malignancy (Gao-2016). One of the reasons is that biomarker and translational research, a prerequisite for the clinically successful disease management, is still in child's shoes in PeCa as compared to many other malignancies. Indeed, fundraising for preclinical research in this condition is challenging and often only possible when applying for funding exclusively dedicated to rare cancers hampering clinical advances as well. In addition, this orphan disease is not "appealing" for drug development pipeline of the pharmaceutical industry due to its rarity in the Western world (Taruscio-2011).

Beside aforementioned aspects, another well-known conundrum - a non-adherence of treating physicians to guideline recommendations - poses a threat to optimization of outcomes in PeCa since available evidence is often only insufficiently utilized in the routine care. A recent survey on local therapy of Tis, Ta-T1a, and T1b PeCa by the European PROspective Penile Cancer Study Group Survey (E-PROPS) distributed across 681 urologists yielded a disenchanted 42.4% adherence rate with a guideline-conform treatment across all tumor stages (Pallauf-2020). A survey assessment in German-speaking countries performed by the same group demonstrated that only 35.2% and 23.9% of 557 participating urologists correctly identified criteria for inguinal and pelvic lymphadenectomy (ILAD, PLAD), respectively (Suarez-Ibarrola-2021). These results are further substantiated by an analysis of the Surveillance, Epidemiology, and End Results and the National Inpatient Sample databases reporting on 24.7% adherence rate with guideline recommendations on ILAD in PeCa (Mistretta-2019). Of note, a recent study using data of 1,689 men diagnosed with pT1b-T3, cN0 PeCa included in the National Cancer Database revealed that only 25.3% of them were subjected to ILAD, omission of which turned out to be an independent predictor of overall mortality (Woldu-2018). This finding underscores the exceptional importance of the appropriate lymph node management in PeCa.

Accordingly, the most decisive prognostic factor for survival in males with PeCa is the presence and extent of nodal metastases, with a 5-year disease-specific survival of approximately 95%, 80%, 65% and 35% for N0, N1, N2 or N3 disease, respectively (Horenblas-1994, Ravi-1993, Wen-2018, Srinivas-1987). Thus, initial lymph node staging is aimed at identifying lymphatic metastasis as early as possible, since superior outcomes have been reported for men with T2-3 cN0 disease at high risk for (micro)metastases subjected to early (prophylactic) as compared to late (therapeutic) ILAD when groin metastases became clinically evident (Kroon-2005). In fact, systemic spread of PeCa occurs in a stepwise manner through the lymphatic system: initially to the inguinal nodes, followed by the pelvic nodes and finally to the retroperitoneal nodes and distant sites, while hematogenic metastasis is rare (Wood-2010, Lopes-1996). Superficial inguinal nodes located in femoral triangle are first affected during dissemination process. Daseler and coworkers divided the superficial inguinal lymph nodes into five regions centered around the saphenofemoral junction; central, lateral superior, lateral inferior, medial superior and medial inferior (Daseler-1948). Hereby, medial superior zone followed by the central inguinal zones contain sentinel inguinal nodes, i.e., those first affected by lymphatic spread (Daseler-1948, Leijte-2008, Omorphos-2018). From superficial lymph nodes further dissemination takes place into deep inguinal nodes located within the region of the fossa ovalis at the saphenofemoral junction as well as medially to the femoral vein up to the node of Cloquet that is located between the femoral vein and the lacunar ligament and marks the most cephalad inguinal lymph node connecting inguinal and iliac/pelvic lymphatics.

If no suspicious nodes are present at palpation (cN0 disease), approximately 20-25% of patients with PeCa may still harbor occult metastases necessitating further risk-adapted staging procedures (Woldu-2018). By now, no validated tumor markers or nomograms are available to predict lymphatic dissemination in PeCa. Since imaging modalities like CT, MRI or 8FDG-PET do not reliably detect metastases < 10 mm, they are not generally recommended in cN0 PeCa, in which the focus is directed at detection of the micrometastatic disease (Jakobsen-2021, Sadeghi-2012). Consequently, surgical staging still maintains its role as the standard care for detection of subclinical metastasis. Due to the morbidity of this strategy, risk categories are used to reduce potential overtreatment for up to 80% of males with cN0 PeCa being free of micrometastatic disease. Well-differentiated (G1), pTa, pTis and pT1 tumours without lymphovascular/perineural invasion and not poorly differentiated (pT1a) are considered low-risk tumours with a neglectable probability of metastases rendering invasive staging unnecessary. Moderately differentiated (G2) pT1a tumors are considered intermediate-risk and are associated with a 6-8% probability of (micro)-metastatic lymph node disease, whereas in pT1b G2 tumors, the risk is 22-30% (Fankhauser-2022). Therefore, all tumors that are stage T1b, or higher, are considered high-risk tumors bearing an up to 80% risk of occult metastasis (Chaux-2015, Solsona-2001). Considering these probabilities, current European Association of Urology (EAU) and American Society of Clinical Oncology (ASCO) Collaborative Guidelines on Penile Cancer recommend surgical lymph node staging for all patients at high risk, while for men at intermediate risk both surgical staging and surveillance with a strict follow-up represent acceptable disease management options (EAU-ASCO Penile Cancer Guidelines). National Comprehensive Cancer Network (NCCN) Guidelines recommend bilateral ILAD as primary surgical staging even in both intermediate and high risk cN0 disease (NCCN Guidelines Penile Cancer 2023).

In patients with palpable nodes in the groin (cN+ disease), nodal metastases are present in approximately 45-80% of cases (Hughes-2009, Lutzen-2016). Notably, for pN1 disease ILAD has been demonstrated to yield similar outcomes as patients with pN0 disease (Martin-2012). Since cure can be achieved in limited lymph node positive disease confined to the regional nodes, radical ILAD is the treatment of choice for males with cN1-2 disease (Brouwer-2023).

The present study is a prospective, investigator-initiated, randomized, open-label phase II trial. Male patients with a histologically proven diagnosis of PeCa and either pT1a G2 cN0, pT1b-3 any G cN0 or pT1-3 any G cN1-2 disease without bulk lymph nodes (< 4cm), constituting the indication for prophylactic or therapeutic inguinal lymphadenectomy, will be enrolled.

The eligible patients will be randomized 1:1 in one of two arms. Patients in the conventional treatment Arm A will receive open inguinal lymphadenectomy and patients in the experimental Arm B will receive robot-assisted inguinal lymphadenectomy. All patients will be followed up for 36 months after last patient in or until death, withdrawal of consent, or loss to follow-up (whichever occurs first).

Investigators will recruit patients directly during regular clinical consultation visits in the respective center. All trial related investigations and enrolment of patients will only be performed after a written informed consent was collected using the ethics committee approved patient information and consent forms.

All patients who gave written informed consent will be captured online in the electronic case report form (eCRF) as screening patients to obtain a patient number which is used for pseudonymized identification throughout the trial.

Provided that all other inclusion and exclusion criteria are met, the patient will be allocated and is allowed to start the trial treatment. If one or more inclusion and/or exclusion criterion is/are not met, the patient will be marked as a screening failure in the eCRF.

Patients will be randomized 1:1 into one of the study arms and stratified by lymph node status (cN0 vs. cN1-2) and body mass index (< 25 vs. ≥ 25). Randomization will be conducted following the allocation by an adaptive randomization procedure implemented in the EDC system.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient has provided written informed consent.
* 2. Male patient ≥ 18 years at time of signing the informed consent form.
* 3. Patient has histologically proven penile squamous cell carcinoma.
* 4. Patient has indication for prophylactic (intermediate or high-risk primary tumor and cN0) or therapeutic (cN1/2) inguinal lymphadenectomy, i.e.:

  * pT1a, G2, cN0 OR
  * pT1b- pT3, any G, cN0 OR
  * pT1-pT3, any G, cN1-2
* 5. Patients has adequate hepatic, renal and bone marrow function:

  * Hemoglobin ≥ 8.0 g/dL
  * Absolute neutrophil count ≥ 1.5 x 109 /L
  * Platelets ≥ 100 x 109 /L
  * International normalized ratio (INR) / activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN unless participant is receiving anticoagulant therapy as long as PTT is within therapeutic range of intended use of anticoagulants. Anticoagulation is accepted according to the surgeon's practice.
* 6. Patient is willing and able to comply with the protocol for the duration of the study, including hospital visits for treatment and scheduled follow-up visits and examinations.
* 7. Performance status of the patient is judged by the treating physician as appropriate to undergo surgery.

Exclusion Criteria:

* 1. Patients has inguinal bulky disease ≥ 4 cm (determined by ultrasound or cross-sectional imaging).
* 2. Patient has distant metastases.
* 3. Patient receives or is scheduled for neoadjuvant chemotherapy for PeCa.
* 4. Patient received previous major inguinal surgery (transabdominal laparoscopic inguinal hernia repair is permitted), lymph node resection or radiotherapy in the groin or pelvic area.
* 5. Patient participates in competing trials affecting the effects of the surgery or outcome measures.
* 6. Patient has addictive or other medical conditions that do not allow the subject to appreciate the nature and scope of the clinical trial and its potential consequences.
* 7. Patient has any co-existing medical condition that in the investigator's judgement will substantially increase the risk associated with the patient's participation in the study.
* 8. Patient has been incarcerated or involuntarily institutionalized by court order or by the authorities.
* 9. Patient is unable to consent because he does not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2026-01-29 (Estimated); Primary Completion 2031-09-30 (Estimated); Study Completion 2031-11-30 (Estimated)

PRIMARY OUTCOMES:
Rate of postoperative complications ≥ grade 3 within 3 months after surgery | Up to 3 months
  Rate of postoperative complications ≥ grade 3 within 3 months after surgery according to Clavien-Dindo classification (Dindo-2004)

SECONDARY OUTCOMES:
Total complication rate | Up to 6 months
  Total complication rate, defined as rate of all post-operative complications that occurred within 4 weeks, 3 and 6 months post-surgery
Drain-free rate | Up to 35 days
  Drain-free rate on day 21, day 28 and day 35 after surgery (drain removal if output < 30 mL/d on at least 3 consecutive days), defined as proportion of patients who no longer have a drain on day 21, 28 and 35 after surgery
Length of drain in situ | Up to drain removal, an average of 3 weeks
  Length of drain in situ, defined as time from surgery to the day of drain removal
Percentage of patients with surgical site infections requiring antibiotic treatment | Up to 6 months
  Percentage of patients with surgical site infections requiring antibiotic treatment
Re-admission rate | Up to 6 months
  Re-admission rate, defined as percentage of admitted patients who return to the hospital for inpatient treatment within 4 weeks, 3 months and 6 months of discharge
Re-operation rate | Up to 5.5 years
  Re-operation rate, defined as percentage of patients with the need for a re-surgery due to complications related to the initial surgery (tumor progress in the groin necessitating further surgical procedures is not counted as an event for the definition "Re-operation rate").
Number of resected lymph nodes per groin and per patient | Day of surgery
  Number of resected lymph nodes per groin and per patient.
Regional recurrence rate | Up to 24 months
  Regional recurrence rate at 12 and 24 months in the groin, defined as proportion of patients with tumor recurrence in the groin at 12 and 24 months after surgery
Regional recurrence-free survival (in the groin) | Up to 5.5 years
  Regional recurrence-free survival (in the groin), defined as time from surgery until the date of recurrence of PeCa in the groin or death from any cause
Metastasis-free survival | Up to 5.5 years
  Metastasis-free survival, defined as time from surgery until the date of spreading of the PeCa to other parts of the body than penis or death from any cause
Disease-free survival | Up to 5.5 years
  Disease-free survival, defined as time from surgery until the date of recurrence of PeCa or death from any cause
Disease-specific survival | Up to 5.5 years
  Disease-specific survival, defined as time from randomization until the date of death from PeCa
Overall survival | Up to 5.5 years
  Overall survival, defined as time from randomization until the date of death from any cause
Local recurrence rate | Up to 5.5 years
  Local recurrence rate (recurrence at penis stump [if initially penis-sparing approach of the primary tumor resection] or adjacent skin [if initially complete penectomy] - independent of the technique of the inguinal lymphadenectomy), defined as proportion of patients with local recurrence of PeCa
General Health-related Quality of Life | Up to 12 months
  General HRQoL: EQ-5D-5L as well as experimental EQ-5D-5L modules (bolt-ons) added to the core measure to address specific concerns for this patient group
Health-related well-being | Up to 12 months
  Health-related well-being: EuroQol Health and Well-Being short-form (EQ-HWB-9)
Quality of recovery from surgery | Up to 12 months
  Quality of recovery from surgery: Postoperative Quality of Recovery Score (PostopQRS)
Sexual Function | Up to 12 months
  Sexual Function: International Index of Erectile Function-5 (IIEF-5)
Depression | Up to 12 months
  Depression: Patient Health Questionnaire-9 (PHQ-9) and Hospital Anxiety and Depression Scale (HADS)
Pain (BPI questionnaire) | Up to 12 months
  Pain: Brief Pain Inventory (BPI) questionnaire
Lymphedema QoL | Up to 12 months
  Lymphedema: condition-specific QoL measure for lymphoedema of the lower limbs (LYMQOL)
QoL - primary informal caregivers | Up to 12 months
  Caregiver completed EQ-5D-5L
QoL - primary informal caregivers | Up to 12 months
  Caregiver completed EQ-HWB-9
Length of hospital stay | Up to discharge from hospital, an average of 5 days
  Length of hospital stay, defined as time from surgery to discharge from hospital
Duration and intensity of procedure-related analgetic treatment | Up to 6 months
  Duration and intensity of procedure-related analgetic treatment
Time to post-surgery scheduled adjuvant or salvage treatment | Up to 5.5 years
  Time to post-surgery scheduled adjuvant or salvage treatment, defined as time from surgery to subsequent adjuvant or salvage treatment (Note: Subsequent palliative systemic treatment in case of emerging new metastasis is not considered)
Cost-benefit analysis | Up to 5.5 years
  Cost data obtained from hospital accounting departments or national cost databases will be used to evaluate the economic impact of robotic versus open inguinal lymphadenectomy. These data will be linked to clinical variables collected in the eCRF.

CONTACTS AND LOCATIONS:
Overall Officials: Igor Tsaur, Prof. Dr., Study Chair — University Hospital Tuebingen, Medical Faculty, Eberhard-Karls-University; Igor Tsaur, Prof. Dr., Principal Investigator — University Hospital Tuebingen, Medical Faculty, Eberhard-Karls-University
Locations (9):
- Germany (9):
  - Charité- Universitätsmedizin Berlin, Berlin
  - University Hospital Carl Gustav Carus, Dresden
  - Universitätsklinikum Erlangen, Erlangen
  - University Medical Center of Johannes Gutenberg-University, Mainz
  - Medical Faculty Mannheim, Mannheim
  - Ludwig Maximilian University Hospital, München
  - University Medicine Rostock, Rostock
  - University Hospital Tübingen, Tübingen
  - University Hospital Ulm, Ulm